CLINICAL TRIAL: NCT06365775
Title: Multi-omics Characteristics and Prognosis in Patients With Idiopathic Sudden Sensorineural Hearing Loss
Brief Title: Multi-omics Characteristics and Prognosis of Idiopathic Sudden Sensorineural Hearing Loss
Status: Not yet recruiting | Type: Observational
Sponsor: Dan Bing (Other)
Responsible Party: Sponsor-Investigator, Dan Bing, associate professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB20221229
Record Dates: First submitted 2023-11-21; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Sudden Sensorineural Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss, Sudden
MeSH Terms: conditions — Hearing Loss, Sudden; Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral venous blood sample.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bilateral SSNHL: 150 participants will be enrolled with SSNHL involving bilateral ears.
- Unilateral SSNHL: 150 participants will be enrolled with SSNHL involving unilateral ear.
- Healthy Controls: 100 age-matched healthy controls will be enrolled.

SUMMARY:
The goal of this observational study is to describe the multi-omics characteristics and to learn about the prognostic factors in patients with idiopathic sudden sensorineural hearing loss (SSNHL). The main problems it aims to deal with are:

* if there is a difference in data of exome and targeted sequencing among patients with SSNHL affecting bilateral and unilateral sides, and healthy controls
* if there is a difference in the parameter of MRI among patients with SSNHL affecting bilateral and unilateral sides, and healthy controls
* to find out which factor from multi-omics data relates to outcomes of SSNHL
* to develop the best prognostics model based on the multi-omics data.

Participants will be received audiological tests, blood specimen collection and radiological examination. Researchers will explore the relationship between the multi-omics data and the prognosis and develop the predictive model.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 4
* Participants with SSNHL: unilateral or bilateral sensorineural hearing loss of > 30 dB HL (decibel) involving at least 3 continuous test frequencies developing within 72 hours
* Healthy controls: people with PTA thresholds of all test frequencies ≤ 20 dB HL and without otologic disease in the last 3 months
* Completed informed consent and promised to finish follow-ups

Exclusion Criteria:

* Hearing loss with explicit causes, including noise-induced, Ménière's disease, ototoxicity exposure, mumps infection or history of syphilis infection and so on.
* A history of head trauma or otologic surgery.
* Malformation of temporal bone discovered by computed tomography (CT)
* Retro-cochlear lesion discovered by magnetic resonance imaging (MRI)
* Pregnant women

Ages: 4 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with SSNHL will be selected from patients diagnosed and treated at Tongji hospital. Participants in healthy controls will be recruited in public from the residents of Wuhan city, China.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-04-23 (Estimated); Primary Completion 2026-11-23 (Estimated); Study Completion 2026-11-23 (Estimated)

PRIMARY OUTCOMES:
Pure tone audiometry (PTA) | Baseline, 14 days, 1, 3 and 6 months follow-ups
  Pure tone thresholds of 250, 500, 1000, 2000, 4000, 8000 Hz will be measured.

SECONDARY OUTCOMES:
Speech reception thresholds | Baseline, 14 days, 1, 3 and 6 months follow-ups
  Speech Reception Thresholds (SRTs) are employed as a critical outcome measure in clinical trials to assess the lowest level at which speech can be understood. This metric is pivotal for evaluating the efficacy of interventions aimed at improving auditory capabilities or mitigating hearing impairments. SRTs are determined through standardized tests where subjects are required to recognize and repeat spoken words or phrases presented at varying volume levels. The threshold is identified as the minimum intensity at which speech is correctly understood 50% of the time. This quantifiable measure allows for the objective comparison of hearing function before and after interventions, making it a valuable tool in clinical research focused on auditory health and rehabilitation.
Speech discrimination scores | Baseline, 14 days, 1, 3 and 6 months follow-ups
  Speech Discrimination Scores (SDS) are a measure used to assess an individual's ability to correctly understand and repeat spoken words. Unlike Speech Reception Thresholds, which focus on the lowest level of audibility, SDS evaluates the clarity of speech understanding at a comfortable listening level. In clinical settings, a list of phonetically balanced words is presented to the participant at a volume that is easily audible, usually set above their speech reception threshold. The score is calculated based on the percentage of words correctly repeated back by the individual. High SDS indicates good speech clarity recognition, while lower scores may suggest difficulties in speech processing or hearing impairments. SDS is crucial in diagnosing, managing, and treating hearing disorders, providing valuable insights into the functional impact of hearing loss and the effectiveness of auditory rehabilitation strategies.

OTHER OUTCOMES:
Variant detection efficiency | Baseline
  The efficiency with which known genetic variants are identified within the targeted regions through capture sequencing of peripheral venous blood samples. This is measured separately for cases and control participants and reported as a percentage (%).
Exome coverage | Baseline
  The extent of coverage achieved in the exome regions within peripheral venous blood samples from cases and controls, quantified by the percentage of the exome sequenced at sufficient depth in whole exome sequencing. Results are reported as a percentage (%) for both groups.
Genome-wide variant distribution | Baseline
  The distribution and density of genetic variants detected across the entire genome in whole genome sequencing of peripheral venous blood samples. This measure is evaluated for both cases and controls and expressed as the number of variants per megabase (variants/Mb).
Head MRI | Baseline
  Assess the integrity of brain tissues, looking for signs of lesions, tumors, or atrophy. This involves qualitative assessments (e.g., presence or absence of abnormalities).
Inner Ear MRI | Baseline
  Detailed assessment of the cochlea and vestibular system's anatomy for structural abnormalities, using a qualitative assessment.